CLINICAL TRIAL: NCT04257890
Title: A Randomized Controlled Trial for Evaluating the Efficacy of a Cognitive Behavioral Therapy Intervention in Reducing Internet Gaming Disorder Among Secondary School Students in Hong Kong
Brief Title: A Cognitive Behavioral Therapy Intervention for Internet Gaming Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Xue YANG, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14607319
Record Dates: First submitted 2019-12-27; First posted 2020-02-06 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT intervention group (Experimental): In addition to the information about IGD of the control group, the intervention group will receive eight weekly group-based 90-minute CBT sessions.
  Interventions: Behavioral: Cognitive behavioral therapy; Other: Education material about IGD; Other: Education material about CBT
- Wait-list control group (Active Comparator): Members will receive printed education material about IGD but not CBT during the treatment period.
  Interventions: Behavioral: Cognitive behavioral therapy; Other: Education material about IGD; Other: Education material about CBT

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — The CBT focuses on cognitive restructuring to reduce the specific key maladaptive beliefs on Internet gaming suggested by King's model, and develop useful coping skills (self-regulation/control, emotion regulation, problem-solving coping) that are adapted from previous CBT for adolescent IGD. In addition, it provides training on relapse-prevention and maintenance techniques.
Other: Education material about IGD — Printed education material introducing IGD will be distributed.
Other: Education material about CBT — Printed education material introducing CBT will be distributed.

SUMMARY:
This RCT study develops a brief group-based CBT intervention. The primary objective is to evaluate the efficacy of the CBT in reducing IGD, compare to a wait-list control group.

DETAILED DESCRIPTION:
Introduction Cognitive behavioral therapy (CBT) is potentially useful as it is effective in treating mental/behavioral disorders, restructuring cognitions and cultivating positive coping. A gap exists as the only two existing clinic-based small randomized controlled trials (RCT) yielded mixed findings on CBT's treatment effect for adolescent IGD.

Objectives This RCT study develops a brief group-based CBT intervention. The primary objective is to evaluate the efficacy of the CBT in reducing IGD, compare to a wait-list control group.

Subjects and methods The study design is two-armed RCT. The participants are Secondary 1-4 students (n=226) with IGD (DSM-5 classification) identified in a school-based screening. Evaluation involves surveys at baseline, end of CBT intervention, and 6 months afterwards. In addition to information received by the wait-list control group, the intervention group receives a carefully designed brief 8-week group-based CBT. The control group will receive CBT after the 6-month follow-up. Trained social workers of a collaborating NGO that serves secondary school students will conduct the CBT.

Outcomes and measures The primary outcome is IGD (a validated DSM-5 IGD classification tool). Secondary outcomes include time spent on Internet/Internet games and the intention to reduce IGD. Measures of potential mediators (maladaptive beliefs and coping) include: Internet Gaming Cognition Scale, Generalized Problematic Internet Use Scale, Emotion Regulation Questionnaire, and Coping Scale for Children and Youth.

Data analysis Intention-to-treat analysis is performed. The primary outcome is assessed by absolute and relative risk reduction. Generalized Linear Mixed Models and Structural Equation Models are used to test secondary outcomes and mediation effects.

Implications The findings may lead to an evidence-based treatment for adolescent IGD, a newly defined disease, which has been rarely reported in literature. Understanding its mechanism contributes to theoretical development of IGD and related treatment.

ELIGIBILITY:
Inclusion Criteria:

* secondary 1-4 students (grade 7-10),
* positive screening results (i.e. IGD cases) according to a validated questionnaire (the 5 DSM-5 criteria for IGD),
* students' and parental consent,
* Chinese speaking.

Exclusion Criteria:

* self-reported history of any psychiatric or neurological illness,
* current use of any psychotropic medication.

We do not include Secondary 5-6 students due to their preparation for public examinations and practical difficulty in follow-up after their graduation.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 226 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Internet gaming disorder (IGD) immediately after the interventions | immediately after the interventions
  The DSM-5 classification of IGD: The 9-item IGD checklist is a short, user-friendly, self-report measure for assessing the DSM-5 classification of IGD. Symptoms to be assessed include preoccupation, tolerance, withdrawal, unsuccessful attempts to limit gaming, deception or lies about gaming, loss of interest in other activities, use despite knowledge of harm, use for escape or relief of negative mood, and harm in the past 12 months. Response options are no (0) and yes (1). As per the DSM-5 recommendation, those with >=5 'yes' responses are considered IGD cases. The Chinese version has been validated with high internal consistency.
Change from baseline Internet gaming disorder (IGD) at 6 months | six months after the interventions
  The DSM-5 classification of IGD: The 9-item IGD checklist is a short, user-friendly, self-report measure for assessing the DSM-5 classification of IGD. Symptoms to be assessed include preoccupation, tolerance, withdrawal, unsuccessful attempts to limit gaming, deception or lies about gaming, loss of interest in other activities, use despite knowledge of harm, use for escape or relief of negative mood, and harm in the past 12 months. Response options are no (0) and yes (1). As per the DSM-5 recommendation, those with >=5 'yes' responses are considered IGD cases. The Chinese version has been validated with high internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yang, Principal Investigator — JC School of Public Health and Primary Care, Faculty of Medicine, CUHK
Locations (6):
- HKMLC Queen Maud Secondary School, Hong Kong, Hong Kong, China
- Hong Kong (5):
  - Henrietta Secondary School, Hong Kong
  - Po Kok Secondary School, Hong Kong
  - Po Leung Kuk Lee Shing Pik College, Hong Kong
  - S.T.F.A. Lee Shau Kee College, Hong Kong
  - Shun Tak Fraternal Association Leung Kau Kui College, Hong Kong

IPD SHARING:
Plan to Share IPD: No